CLINICAL TRIAL: NCT05547217
Title: Gamification of Neurorehabilitation-centric Hand Exercises Post Stroke or Brain Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRegained Inc. (Industry)
Collaborators: Laurentian University, Health Science North (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUSUON0002
Record Dates: First submitted 2022-09-14; First posted 2022-09-21 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Engagement, Patient
MeSH Terms: conditions — Stroke; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurorehabilitation of the Hand (Experimental): Participants will undergo a 2-hour training session, 2-3 days per week, over 12 weeks, for a total of 30 sessions. Hand function therapy will be administered in a specific and gamified manner to enhance rehabilitation of the hand and provide participants with greater opportunity to regain hand function over the course of the study.
  Interventions: Device: Hand Therapy using the MyHand System

INTERVENTIONS:
Device: Hand Therapy using the MyHand System — The MyHandTM System is a smart-mechatronic device programmed with proprietary hand function training regiments (protocols) based on deep research in neuroplasticity. It provides a highly unique and targeted approach to hand function rehabilitation with the help of the aforementioned protocols delivered with gamified training techniques. The gamified format of the protocols allows for better patient engagement, thus allowing for more effective and efficient therapy. Participants will undergo a 2-hour training session, 2-3 days per week, over 12 weeks, for a total of 30 sessions. Hand function therapy will be administered in a specific and gamified manner to enhance rehabilitation of the hand and provide participants with greater opportunity to regain hand function over the course of the study.

SUMMARY:
Stroke is the leading cause of adult disability worldwide. Often, severe neurological deficits occur after a stroke and roughly 70% of all stroke survivors have some form of hand function disability. To improve the lives of those with hand function disability, IRegained Inc. has created the MyHandTM System. The MyHandTM System is a smart-mechatronic device programmed with proprietary hand function training regiments (protocols) based on deep research in neuroplasticity. It provides a highly unique and targeted approach to hand function rehabilitation with the help of the aforementioned protocols delivered with gamified training techniques. The gamified format of the protocols allows for better patient engagement, thus allowing for more effective and efficient therapy. Individuals who have sustained a stroke 5 months or earlier (considered to be chronic stroke survivors) will be eligible to participate in this study. Participants will undergo a 2-hour training session, 2-3 days per week, over 12 weeks, for a total of 30 sessions. Hand function therapy will be administered in a specific and gamified manner to enhance rehabilitation of the hand and provide participants with greater opportunity to regain hand function over the course of the study. The goal of this research project is to understand how a gamified approach to hand function rehabilitation impacts engagement and motivation. This understanding will directly translate into the development of more efficient and effective modes of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a single stroke

Exclusion Criteria:

* Severe spasticity or contractures (2 or less in the CMSA) or any other musculoskeletal or neuromuscular disorders that compromise sensation or other neuromuscular parameters will be excluded from the study. Prospective participants who are incapable of providing consent to participate in the research study will also be excluded (determined by an MMSE score of 23 or less).

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-09-19 (Estimated); Study Completion 2023-09-19 (Estimated)

PRIMARY OUTCOMES:
the Chedoke Arm and Hand Activity Inventory -9 (CAHAI-9)- Change is being assessed | Baseline- before beginning the treatment, INTRA- after the completion of 15 treatment sessions and Post treatment- after the conclusion of 30 treatment sessions
  a 9-item assessment, will be performed by a trained clinician to estimate a participants functional ability during the initial assessment. The CAHAI-9 requires a participant to perform 9 bimanual ADLs, each of which will be scored on a 7 point scale.
Box and Block Test- Change is being assessed | Baseline- before beginning the treatment, INTRA- after the completion of 15 treatment sessions and Post treatment- after the conclusion of 30 treatment sessions
  The BBT requires participants to move cubical wooden blocks over a partition from one box to another. Grip and pinch dynamometry will be used to assess a participant's hand strength.
The Motor Activity Log- Change is being assessed | Baseline- before beginning the treatment, INTRA- after the completion of 15 treatment sessions and Post treatment- after the conclusion of 30 treatment sessions
  Estimates how much and how well a participant is able to use their affected upper limb. The MAL is a 30 item questionnaire administered in through a semi-structured interview between the participant and a trained clinician.
the NASA-Task Load Index (NASA-TLX)- Change is being assessed | After each treatment session
  an assessment tool used to evaluate a participants perceived cognitive load during a session. The NASA-TLX has six sub-scales; mental demand, temporal demand, frustration, performance, effort and physical demand. The NASA-TLX scores, time taken to complete a level, game score and verbal language references made during gameplay will be used to estimate engagement.
European Quality of Life Five Dimension Questionnaire (EQ-5D)- Change is being assessed | Baseline- before beginning the treatment and Post treatment- after the conclusion of 30 treatment sessions
  To measure participants perceived quality of life through a questionnaire.

SECONDARY OUTCOMES:
Finger Goniometry- Change is being assessed | Baseline- before beginning the treatment, INTRA- after the completion of 15 treatment sessions and Post treatment- after the conclusion of 30 treatment sessions
  estimate range of motion (ROM) of the various finger joints.
Grip Dynamometry- Change is being assessed | Baseline- before beginning the treatment, INTRA- after the completion of 15 treatment sessions and Post treatment- after the conclusion of 30 treatment sessions
  Measures participants grip strength
Pinch Dynamometry- Change is being assessed | Baseline- before beginning the treatment, INTRA- after the completion of 15 treatment sessions and Post treatment- after the conclusion of 30 treatment sessions
  Measures participants pinch strength

CONTACTS AND LOCATIONS:
Locations (1):
- Laurentian University, Greater Sudbury, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No